CLINICAL TRIAL: NCT02186847
Title: Randomized Phase II Trial of Concurrent Chemoradiotherapy +/- Metformin HCL in Locally Advanced NSCLC
Brief Title: Chemotherapy and Radiation Therapy With or Without Metformin Hydrochloride in Treating Patients With Stage III Non-small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: NRG Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NRG-LU001; NCI-2014-01071 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); PNRG-LU001_A01PAMDREVW01; NRG-LU001 (Other: NRG Oncology); NRG-LU001 (Other: CTEP); U10CA180868 (NIH)
Record Dates: First submitted 2014-07-08; First posted 2014-07-10 (Estimated); Results first posted 2020-06-23 (Actual); Last update posted 2025-10-09 (Actual); Status verified 2025-09

CONDITIONS: Adenosquamous Lung Carcinoma; Bronchioloalveolar Carcinoma; Large Cell Lung Carcinoma; Lung Adenocarcinoma; Non-Small Cell Lung Carcinoma; Recurrent Non-Small Cell Lung Carcinoma; Squamous Cell Lung Carcinoma; Stage IIIA Non-Small Cell Lung Cancer; Stage IIIB Non-Small Cell Lung Cancer
MeSH Terms: conditions — Adenocarcinoma, Bronchiolo-Alveolar; Adenocarcinoma of Lung; Carcinoma, Non-Small-Cell Lung | interventions — Radiotherapy; Radiotherapy, Conformal; Radiotherapy, Intensity-Modulated; Carboplatin; Metformin; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Chemoradiation (Active Comparator): 60 Gy Radiation therapy with concurrent paclitaxel and carboplatin followed by consolidation paclitaxel and carboplatin
  Interventions: Radiation: Radiation Therapy; Drug: Carboplatin; Drug: Paclitaxel
- Metformin + Chemoradiation (Experimental): Metformin plus 60 Gy Radiation therapy with concurrent paclitaxel and carboplatin followed by consolidation paclitaxel and carboplatin
  Interventions: Radiation: Radiation Therapy; Drug: Carboplatin; Drug: Metformin; Drug: Paclitaxel

INTERVENTIONS:
Radiation: Radiation Therapy — Radiation therapy (RT) is given in 2 Gy fractions once daily 5 days per week to a total of 30 fractions and 60 Gy. Photons required; 3-dimensional conformal radiation therapy (3D-CRT) or intensity-modulated radiation therapy (IMRT) permitted. Starts within 14 days of randomization (Chemoradiation arm) or 14 days after metformin starts (Chemoradiation + Metformin arm).
  Other Names: 3-dimensional conformal radiation therapy; 3D-CRT; Intensity-modulated radiation therapy; IMRT
Drug: Carboplatin — 2 AUC (area under the curve) via IV weekly on days 1, 8, 15, 22, 29, and 36 from start of radiation therapy. Two 21 day cycles of 6 AUC via IV starting 28-42 days after the end of radiation therapy.
Drug: Metformin — Metformin is taken orally. Dose escalation begins 2 weeks prior to the initiation of chemoradiation. 500 mg twice daily days 1-7 of metformin. 500 mg three times daily days 8-14 of metformin. Three times a day with the following dosage: 500mg in the morning, 1000mg at noon, and 500mg in the evening concurrent with chemoradiation and through consolidation chemotherapy (days 15-126 of metformin),
  Other Names: Metformin HCL; Metformin Hydrochloride
  Arms: Metformin + Chemoradiation
Drug: Paclitaxel — 50 mg/m2 via IV weekly on days 1, 8, 15, 22, 29, and 36 from start of radiation therapy. Two 21 day cycles of 200 mg/m2 via IV 28-42 days after the end of radiation therapy.

SUMMARY:
This randomized phase II trial studies how well chemotherapy and radiation therapy given with or without metformin hydrochloride works in treating patients with stage III non-small cell lung cancer. Drugs used in chemotherapy, such as carboplatin and paclitaxel, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Radiation therapy uses high-energy x-rays to kill tumor cells and shrink tumors. Metformin hydrochloride may shrink tumors and keep them from coming back. It is not yet known whether chemotherapy and radiation therapy is more effective when given with or without metformin hydrochloride in treating stage III non-small cell lung cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine whether metformin hydrochloride (MET) added to chemoradiotherapy can improve progression-free survival (PFS) in patients with locally advanced non-small cell lung cancer (NSCLC).

SECONDARY OBJECTIVES:

I. Determine the effects of MET on overall survival (OS), time to local-regional progression (LRP), and time to distant metastasis (DM).

II. Evaluate the effect of MET on chemoradiotherapy toxicity (Common Terminology Criteria for Adverse Events, version 4 [CTCAE, v. 4]) within 1 year of completion of all treatment.

III. Collect biospecimens to develop biomarkers of MET activity.

OUTLINE: Patients are randomized to 1 of 2 treatment arms.

After completion of study treatment, patients are followed up at 4-6 weeks, every 3 months for 2 years, every 6 months for 3 years, and then annually thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically (histologically or cytologically) proven diagnosis of stage IIIA or IIIB non-small cell lung cancer within 84 days of registration; eligible histologies include adenocarcinoma, adenosquamous, large cell carcinoma, squamous carcinoma, non-lobar and non-diffuse bronchoalveolar cell carcinoma or non-small cell lung cancer not otherwise specified)
* Patients must have measurable disease
* Patients must have unresectable disease, be medically inoperable, or unwilling to undergo surgical management
* Appropriate stage for protocol entry, including no distant metastases, based upon the following minimum diagnostic workup:

  * History/physical examination, including documentation of height, weight, body surface area, and vital signs, within 30 days prior to registration
  * Computed tomography (CT) with IV contrast or magnetic resonance imaging (MRI) imaging (if CT scan with contrast is medically contraindicated) of the lung and upper abdomen through the adrenal glands, required within 45 days prior to registration (recommended within 30 days prior to registration
  * MRI of the brain with contrast (or CT with contrast if MRI is medically contraindicated) within 45 days prior to registration; note: the use of intravenous contrast is required for the MRI or CT; an MRI without contrast is only permitted if the patient has a contrast allergy
  * Whole-body fludeoxyglucose (FDG)-positron emission tomography (PET)/CT required within 45 days prior to registration (recommended within 30 days prior to registration; note: patients do not need to have a separate CT of the chest and upper abdomen with contrast if PET/CT imaging includes a high quality CT with contrast
* Zubrod performance status 0-1
* Absolute neutrophil count (ANC) >= 1,500 cells/mm^3
* Complete blood count(CBC)/differential obtained within 14 days prior to registration on study, with adequate bone marrow function defined as follows:

  * Absolute neutrophil count (ANC) ≥ 1,500 cells/mm3
  * Platelets >= 100,000 cells/mm^3
  * Hemoglobin >= 8.0 g/dl (note: the use of transfusion or other intervention to achieve hemoglobin [Hgb] >= 8.0 g/dl is acceptable)
* Adequate renal function within 14 days prior to registration, defined as serum creatinine within normal institutional limits or creatinine clearance must be at least 60 ml/min;
* Adequate hepatic function within 14 days prior to registration, defined as total bilirubin ≤ 1.5 x upper limit of normal (ULN) for the institution and alanine aminotransferase (ALT), aspartate aminotransferase (AST), and alkaline phosphatase ≤ 2.5 x ULN for the institution;
* Fasting blood glucose ≤ 125 mg/dL within 14 days prior to registration;
* Serum albumin > 3.0 g/dl within 14 days prior to registration;
* For women of childbearing potential, a serum pregnancy test within 72 hours prior to registration;
* Patients with post-obstructive pneumonia are eligible provided they no longer require intravenous antibiotics at registration;
* Patients must be at least 3 weeks from prior thoracotomy (if performed);
* If a pleural effusion is present, the following criteria must be met at registration to exclude malignant involvement (incurable M1a disease):

  * When pleural fluid is visible on both the CT scan and on a chest x-ray, a pleuracentesis is required to confirm that the pleural fluid is cytologically negative;
  * Effusions that are minimal (i.e. not visible under ultrasound guidance) and that are too small to safely tap are eligible.
* Women of childbearing potential and male participants must practice adequate contraception throughout the study;

Exclusion Criteria:

* Patients with mixed small cell and non-small cell histologies
* Patients with distant metastasis
* Prior invasive malignancy (except non-melanomatous skin cancer) unless disease free for a minimum of 3 years (for example, carcinoma in situ of the breast, oral cavity, or cervix are all permissible)
* Prior systemic chemotherapy for the study cancer; note that prior chemotherapy for a different cancer is allowable
* Prior radiotherapy to the region of the study cancer that would result in overlap of radiation therapy fields
* Patients currently using metformin (metformin hydrochloride), other oral hypoglycemic agents or insulin
* Patients with any history of allergic reaction to paclitaxel or other taxanes or carboplatin
* Patients with a history of chronic kidney disease or lactic acidosis
* Patients with >= 10% weight loss within the past month
* Severe, active co-morbidity, defined as follows:

  * Diagnosis of type I or type II diabetes mellitus
  * Uncontrolled neuropathy >= grade 2 regardless of cause
  * Unstable angina and/or congestive heart failure requiring hospitalization within the last 6 months
  * Transmural myocardial infarction within the last 6 months
  * Acute bacterial or fungal infection requiring intravenous antibiotics at the time of registration
  * Chronic obstructive pulmonary disease exacerbation or other respiratory illness requiring hospitalization or precluding study therapy within 30 days of registration
  * Severe hepatic disease, defined as a diagnosis of Child-Pugh class B or C hepatic disease
  * Human immunodeficiency virus (HIV) positive with cluster of differentiation (CD)4 count < 200 cells/microliter; note that patients who are HIV positive are eligible, provided they are under treatment with highly active antiretroviral therapy (HAART) and have a CD4 count >= 200 cells/microliter within 30 days prior to registration; note also that HIV testing is not required for eligibility for this protocol
  * End-stage renal disease (ie, on dialysis or dialysis has been recommended)
* Pregnancy or women of childbearing potential and men who are sexually active and not willing/able to use medically acceptable forms of contraception

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Actual)
Dates: Start 2014-08; Primary Completion 2019-04-16 (Actual); Study Completion 2025-09-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Theodoros Tsakiridis, Principal Investigator — NRG Oncology
Locations (224):
- United States (220):
  - Lewis and Faye Manderson Cancer Center, Tuscaloosa, Alabama
  - Banner University Medical Center - Tucson, Tucson, Arizona
  - Sutter Cancer Centers Radiation Oncology Services-Auburn, Auburn, California
  - Sutter Cancer Centers Radiation Oncology Services-Cameron Park, Cameron Park, California
  - Eden Hospital Medical Center, Castro Valley, California
  - UC San Diego Moores Cancer Center, La Jolla, California
  - Memorial Medical Center, Modesto, California
  - Kaiser Permanente Oakland-Broadway, Oakland, California
  - Kaiser Permanente-Rancho Cordova Cancer Center, Rancho Cordova, California
  - Rohnert Park Cancer Center, Rohnert Park, California
  - Sutter Cancer Centers Radiation Oncology Services-Roseville, Roseville, California
  - The Permanente Medical Group-Roseville Radiation Oncology, Roseville, California
  - Sutter Medical Center Sacramento, Sacramento, California
  - South Sacramento Cancer Center, Sacramento, California
  - UCSF Medical Center-Mount Zion, San Francisco, California
  - Kaiser Permanente Cancer Treatment Center, South San Francisco, California
  - Sutter Cancer Centers Radiation Oncology Services-Vacaville, Vacaville, California
  - University of Colorado Hospital, Aurora, Colorado
  - Penrose-Saint Francis Healthcare, Colorado Springs, Colorado
  - UCHealth Memorial Hospital Central, Colorado Springs, Colorado
  - Swedish Medical Center, Englewood, Colorado
  - North Colorado Medical Center, Greeley, Colorado
  - McKee Medical Center, Loveland, Colorado
  - SCL Health Lutheran Medical Center, Wheat Ridge, Colorado
  - Christiana Care Health System-Christiana Hospital, Newark, Delaware
  - UF Cancer Center at Orlando Health, Orlando, Florida
  - 21st Century Oncology-Palatka, Palatka, Florida
  - Piedmont Hospital, Atlanta, Georgia
  - John B Amos Cancer Center, Columbus, Georgia
  - Dekalb Medical Center, Decatur, Georgia
  - Memorial Health University Medical Center, Savannah, Georgia
  - Lewis Cancer and Research Pavilion at Saint Joseph's/Candler, Savannah, Georgia
  - Queen's Medical Center, Honolulu, Hawaii
  - The Cancer Center of Hawaii-Liliha, Honolulu, Hawaii
  - The Cancer Center of Hawaii-Pali Momi, ‘Aiea, Hawaii
  - Saint Alphonsus Cancer Care Center-Boise, Boise, Idaho
  - Kootenai Cancer Center, Post Falls, Idaho
  - Saint Luke's Mountain States Tumor Institute-Twin Falls, Twin Falls, Idaho
  - Northwest Community Hospital, Arlington Heights, Illinois
  - John H Stroger Jr Hospital of Cook County, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Good Samaritan Regional Health Center, Mount Vernon, Illinois
  - OSF Saint Francis Radiation Oncology at Pekin Cancer Treatment Center, Pekin, Illinois
  - OSF Saint Francis Radiation Oncology at Peoria Cancer Center, Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - OSF Saint Francis Medical Center, Peoria, Illinois
  - Memorial Medical Center, Springfield, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - IU Health Bloomington, Bloomington, Indiana
  - Radiation Oncology Associates PC, Fort Wayne, Indiana
  - Parkview Hospital Randallia, Fort Wayne, Indiana
  - Franciscan Health Indianapolis, Indianapolis, Indiana
  - Mercy Hospital, Cedar Rapids, Iowa
  - University of Kansas Cancer Center, Kansas City, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - University of Kansas Cancer Center-Overland Park, Overland Park, Kansas
  - Ascension Via Christi Hospitals Wichita, Wichita, Kansas
  - Wesley Medical Center, Wichita, Kansas
  - Hardin Memorial Hospital, Elizabethtown, Kentucky
  - Baptist Health Lexington, Lexington, Kentucky
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - LSU Health Baton Rouge-North Clinic, Baton Rouge, Louisiana
  - Louisiana Hematology Oncology Associates LLC, Baton Rouge, Louisiana
  - Mary Bird Perkins Cancer Center, Baton Rouge, Louisiana
  - Our Lady of the Lake Physicians Group - Medical Oncology, Baton Rouge, Louisiana
  - Mary Bird Perkins Cancer Center - Covington, Covington, Louisiana
  - Mary Bird Perkins Cancer Center - Houma, Houma, Louisiana
  - Maine Medical Center- Scarborough Campus, Scarborough, Maine
  - University of Maryland/Greenebaum Cancer Center, Baltimore, Maryland
  - UM Upper Chesapeake Medical Center, Bel Air, Maryland
  - UM Baltimore Washington Medical Center/Tate Cancer Center, Glen Burnie, Maryland
  - Peninsula Regional Medical Center, Salisbury, Maryland
  - Boston Medical Center, Boston, Massachusetts
  - Lowell General Hospital, Lowell, Massachusetts
  - Henry Ford Hospital, Detroit, Michigan
  - McLaren Cancer Institute-Flint, Flint, Michigan
  - Mercy Health Saint Mary's, Grand Rapids, Michigan
  - Spectrum Health at Butterworth Campus, Grand Rapids, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - McLaren Cancer Institute-Lapeer Region, Lapeer, Michigan
  - McLaren Cancer Institute-Macomb, Mount Clemens, Michigan
  - McLaren Cancer Institute-Central Michigan, Mount Pleasant, Michigan
  - Mercy Health Mercy Campus, Muskegon, Michigan
  - McLaren Cancer Institute-Owosso, Owosso, Michigan
  - McLaren Cancer Institute-Northern Michigan, Petoskey, Michigan
  - Saint Joseph Mercy Oakland, Pontiac, Michigan
  - William Beaumont Hospital-Royal Oak, Royal Oak, Michigan
  - Lakeland Medical Center Saint Joseph, Saint Joseph, Michigan
  - William Beaumont Hospital - Troy, Troy, Michigan
  - Sanford Joe Lueken Cancer Center, Bemidji, Minnesota
  - Mercy Hospital, Coon Rapids, Minnesota
  - Saint Luke's Hospital of Duluth, Duluth, Minnesota
  - Fairview-Southdale Hospital, Edina, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Rice Memorial Hospital, Willmar, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - Southeast Cancer Center, Cape Girardeau, Missouri
  - North Kansas City Hospital, Kansas City, Missouri
  - The University of Kansas Cancer Center-South, Kansas City, Missouri
  - The University of Kansas Cancer Center-North, Kansas City, Missouri
  - The University of Kansas Cancer Center-Lee's Summit, Lee's Summit, Missouri
  - Delbert Day Cancer Institute at PCRMC, Rolla, Missouri
  - CoxHealth South Hospital, Springfield, Missouri
  - Missouri Baptist Medical Center, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Billings Clinic Cancer Center, Billings, Montana
  - Community Medical Hospital, Missoula, Montana
  - CHI Health Saint Francis, Grand Island, Nebraska
  - CHI Health Good Samaritan, Kearney, Nebraska
  - Nebraska Methodist Hospital, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Wentworth-Douglass Hospital, Dover, New Hampshire
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - Virtua Memorial, Mount Holly, New Jersey
  - Community Medical Center, Toms River, New Jersey
  - Virtua Voorhees, Voorhees Township, New Jersey
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - New Mexico Oncology Hematology Consultants, Albuquerque, New Mexico
  - New York-Presbyterian/Brooklyn Methodist Hospital, Brooklyn, New York
  - University of Rochester, Rochester, New York
  - Gaston Hematology and Oncology Associates-Belmont, Belmont, North Carolina
  - CaroMont Regional Medical Center, Gastonia, North Carolina
  - Gaston Hematology and Oncology Associates, Gastonia, North Carolina
  - FirstHealth of the Carolinas-Moore Regional Hospital, Pinehurst, North Carolina
  - Sanford Bismarck Medical Center, Bismarck, North Dakota
  - Sanford Roger Maris Cancer Center, Fargo, North Dakota
  - UHHS-Chagrin Highlands Medical Center, Beachwood, Ohio
  - Mercy Medical Center, Canton, Ohio
  - Aultman Health Foundation, Canton, Ohio
  - Geauga Hospital, Chardon, Ohio
  - Adena Regional Medical Center, Chillicothe, Ohio
  - University of Cincinnati/Barrett Cancer Center, Cincinnati, Ohio
  - Case Western Reserve University, Cleveland, Ohio
  - Cleveland Clinic Cancer Center/Fairview Hospital, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - The Mark H Zangmeister Center, Columbus, Ohio
  - Mount Carmel Health Center West, Columbus, Ohio
  - Good Samaritan Hospital - Dayton, Dayton, Ohio
  - Mercy Cancer Center-Elyria, Elyria, Ohio
  - Cleveland Clinic Cancer Center Independence, Independence, Ohio
  - Kettering Medical Center, Kettering, Ohio
  - Hillcrest Hospital Cancer Center, Mayfield Heights, Ohio
  - UH Seidman Cancer Center at Lake Health Mentor Campus, Mentor, Ohio
  - UH Seidman Cancer Center at Southwest General Hospital, Middleburg Heights, Ohio
  - Newark Radiation Oncology, Newark, Ohio
  - University Hospitals Parma Medical Center, Parma, Ohio
  - Southern Ohio Medical Center, Portsmouth, Ohio
  - North Coast Cancer Care, Sandusky, Ohio
  - UH Seidman Cancer Center at Firelands Regional Medical Center, Sandusky, Ohio
  - Cleveland Clinic Cancer Center Strongsville, Strongsville, Ohio
  - University Pointe, West Chester, Ohio
  - UHHS-Westlake Medical Center, Westlake, Ohio
  - Cleveland Clinic Wooster Family Health and Surgery Center, Wooster, Ohio
  - Genesis Healthcare System Cancer Care Center, Zanesville, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Abington Memorial Hospital, Abington, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Northeast Radiation Oncology Center, Dunmore, Pennsylvania
  - The Regional Cancer Center, Erie, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - UPMC-Shadyside Hospital, Pittsburgh, Pennsylvania
  - Reading Hospital, West Reading, Pennsylvania
  - Geisinger Wyoming Valley/Henry Cancer Center, Wilkes-Barre, Pennsylvania
  - Lankenau Medical Center, Wynnewood, Pennsylvania
  - AnMed Health Cancer Center, Anderson, South Carolina
  - Greenville Health System Cancer Institute-Faris, Greenville, South Carolina
  - Saint Francis Cancer Center, Greenville, South Carolina
  - Greenville Health System Cancer Institute-Eastside, Greenville, South Carolina
  - Self Regional Healthcare, Greenwood, South Carolina
  - Greenville Health System Cancer Institute-Greer, Greer, South Carolina
  - Gibbs Cancer Center-Pelham, Greer, South Carolina
  - Greenville Health System Cancer Institute-Seneca, Seneca, South Carolina
  - Spartanburg Medical Center, Spartanburg, South Carolina
  - Greenville Health System Cancer Institute-Spartanburg, Spartanburg, South Carolina
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - University of Texas Medical Branch, Galveston, Texas
  - M D Anderson Cancer Center, Houston, Texas
  - The Methodist Hospital System, Houston, Texas
  - MD Anderson in Katy, Houston, Texas
  - UTMB Cancer Center at Victory Lakes, League City, Texas
  - MD Anderson League City, Nassau Bay, Texas
  - MD Anderson in Sugar Land, Sugar Land, Texas
  - MD Anderson in The Woodlands, The Woodlands, Texas
  - Intermountain Medical Center, Murray, Utah
  - Central Vermont Medical Center/National Life Cancer Treatment, Berlin Corners, Vermont
  - University of Vermont Medical Center, Burlington, Vermont
  - Norris Cotton Cancer Center-North, Saint Johnsbury, Vermont
  - Augusta Health Center for Cancer and Blood Disorders, Fishersville, Virginia
  - Harrison Medical Center, Bremerton, Washington
  - PeaceHealth Saint John Medical Center, Longview, Washington
  - PeaceHealth Southwest Medical Center, Vancouver, Washington
  - Wheeling Hospital/Schiffler Cancer Center, Wheeling, West Virginia
  - Aurora Cancer Care-Grafton, Grafton, Wisconsin
  - Aurora BayCare Medical Center, Green Bay, Wisconsin
  - Aurora Cancer Care-Kenosha South, Kenosha, Wisconsin
  - Bay Area Medical Center, Marinette, Wisconsin
  - Marshfield Medical Center-Marshfield, Marshfield, Wisconsin
  - Community Memorial Hospital, Menomonee Falls, Wisconsin
  - Ascension Columbia Saint Mary's Hospital Ozaukee, Mequon, Wisconsin
  - Ascension Columbia Saint Mary's Water Tower Medical Commons, Milwaukee, Wisconsin
  - Aurora Saint Luke's Medical Center, Milwaukee, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
  - Zablocki Veterans Administration Medical Center, Milwaukee, Wisconsin
  - Marshfield Clinic-Minocqua Center, Minocqua, Wisconsin
  - Cancer Center of Western Wisconsin, New Richmond, Wisconsin
  - Marshfield Medical Center-Rice Lake, Rice Lake, Wisconsin
  - Saint Michael's Hospital, Stevens Point, Wisconsin
  - Aurora Medical Center in Summit, Summit, Wisconsin
  - Vince Lombardi Cancer Clinic-Two Rivers, Two Rivers, Wisconsin
  - Aurora West Allis Medical Center, West Allis, Wisconsin
  - The Alyce and Elmore Kraemer Cancer Care Center, West Bend, Wisconsin
  - Diagnostic and Treatment Center, Weston, Wisconsin
  - Aspirus UW Cancer Center, Wisconsin Rapids, Wisconsin
- Canada (3):
  - Jewish General Hospital, Montreal, Quebec
  - Allan Blair Cancer Centre, Regina, Saskatchewan
  - Saskatoon Cancer Centre, Saskatoon, Saskatchewan
- Chaim Sheba Medical Center, Tel Litwinsky, Israel

REFERENCES:
- [Derived] Skinner H, Hu C, Tsakiridis T, Santana-Davila R, Lu B, Erasmus JJ, Doemer AJ, Videtic GMM, Coster J, Yang AX, Lee RY, Werner-Wasik M, Schaner PE, McCormack SE, Esparaz BT, McGarry RC, Bazan J, Struve T, Paulus R, Bradley JD. Addition of Metformin to Concurrent Chemoradiation in Patients With Locally Advanced Non-Small Cell Lung Cancer: The NRG-LU001 Phase 2 Randomized Clinical Trial. JAMA Oncol. 2021 Sep 1;7(9):1324-1332. doi: 10.1001/jamaoncol.2021.2318. PMID 34323922

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Chemoradiation | Metformin + Chemoradiation
Started | 84 | 86
Eligible Population | 81 | 86
Eligible and Started Protocol Treatment | 76 | 82
Completed (Participants contributing data to results are considered to have completed the study.) | 81 | 86
Not Completed | 3 | 0
Not completed — Protocol Violation | 3 | 0

BASELINE CHARACTERISTICS:
Population: Eligible participants
Groups:
- Total: Total of all reporting groups
Arm/Group | Chemoradiation | Metformin + Chemoradiation | Total
Number analyzed (Participants) | 81 | 86 | 167
Age, Customized [Count of Participants; unit: Participants] — years
  Participants
    ≤ 49 | 6 | 3 | 9
    50-59 | 22 | 26 | 48
    60-69 | 29 | 35 | 64
    ≥ 70 | 24 | 22 | 46
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 48 | 49 | 97
  Male | 33 | 37 | 70
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 1 | 4
  Not Hispanic or Latino | 77 | 80 | 157
  Unknown or Not Reported | 1 | 5 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 0 | 2
  Asian | 5 | 2 | 7
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 7 | 7 | 14
  White | 67 | 70 | 137
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 5 | 5
Zubrod performance status [Count of Participants; unit: Participants] — 0 = Asymptomatic; 1 = Symptomatic but completely ambulatory; 2 = Symptomatic, <50% in bed during the day; 3 = Symptomatic, >50% in bed, but not bed bound; 4 = Bedbound; 5 = Death
  Participants
    0 | 38 | 45 | 83
    1 | 43 | 41 | 84
American Joint Committee on Cancer (AJCC ) Stage, 7th edition [Count of Participants; unit: Participants] — Tumor stage refers to the size and/or extent of the main tumor. The higher the number after the T, the larger the tumor or the more it has grown into nearby tissues. T's may be further divided to provide more detail, such as T3a and T3b.TX=Primary tumor not visualized by imaging or bronchoscopy. Regional lymph nodes staging refers to the number and/or extent of spread of lymph nodes that contain cancer. The higher the number after the N, the greater the involvement of regional lymph nodes. M0=No distant metastasis
  Participants
    IIIA (M0:T1a-b,N2;T2a-b,N2;T3,N1-2;T4,N0-1) | 52 | 58 | 110
    IIIB (M0: T1a-b,N3;T2a-b,N3;T3,N3;T4,N2-3) | 28 | 26 | 54
    N2,TX, M0 | 1 | 2 | 3
Histology [Count of Participants; unit: Participants]
  Adenocarcinoma | 31 | 42 | 73
  Adenosquamous | 1 | 0 | 1
  Non-small cell lung cancer NOS | 11 | 9 | 20
  Squamous cell carcinoma | 38 | 35 | 73
Did the patient use cigarettes? [Count of Participants; unit: Participants]
  No | 5 | 6 | 11
  Yes, but quit | 47 | 52 | 99
  Yes, currently smokes | 22 | 20 | 42
  Unknown | 7 | 8 | 15

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Alive Without Progression (Progression-free Survival)
Description: Progression is defined per RECIST v1.1 as change in a known lesion(s) meeting one of the following criteria: [1] At least a 20% increase in the sum of the longest diameter of target lesions such that the absolute increase must be > 5 mm. [2] Appearance of ≥1 new lesions. Progression-free survival time is defined as time from randomization to the date of first progression, death, or last known follow-up (censored). Progression-free survival rates are estimated using the Kaplan-Meier method. The protocol specifies that the distributions of failure times be compared between the arms, which is reported in the statistical analysis results. One-year rates are provided. Analysis occurred after 102 progression-free survival events were reported.
Time Frame: From randomization to last follow-up. Maximum follow-up at time of analysis was 47.2 months.
Population: Eligible participants
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Chemoradiation | Metformin + Chemoradiation
Number analyzed (Participants) | 81 | 86
percentage of participants | 60.4 [48.5 to 70.4] | 51.3 [39.8 to 61.7]
Statistical Analysis 1: Comparison: Chemoradiation vs Metformin + Chemoradiation; The study was powered to detect an improvement of the 1-year progression-free survival rate from 50% (no metformin) to 65% (metformin) or equivalently a hazard ratio (HR) of 0.622, at one-sided type 1 error of 0.1 and 85% power with at least 102 progression-free survival events; Test type: Superiority; p = 0.7563, Log Rank; One-sided significance level = 0.10; Hazard Ratio (HR) = 1.15, 95% CI 2-sided [0.77 to 1.73] — Reference level = Chemoradiation

2. Secondary Outcome: Percentage of Participants Alive (Overall Survival)
Description: Overall survival time is defined as time from randomization to the date of death from any cause or last known follow-up (censored). Overall survival rates are estimated using the Kaplan-Meier method. The protocol specifies that the distributions of failure times be compared between the arms, which is reported in the statistical analysis results. One-year rates are provided. Analysis occurred after 102 progression-free survival events were reported.
Time Frame: From randomization to last follow-up. Maximum follow-up at time of analysis was 47.2 months.
Population: Eligible participants
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Chemoradiation | Metformin + Chemoradiation
Number analyzed (Participants) | 81 | 86
percentage of participants | 38.5 [26.3 to NA] — Not reached | 40.1 [27.9 to NA] — Not reached
Statistical Analysis 1: Comparison: Chemoradiation vs Metformin + Chemoradiation; Test type: Superiority; p = 0.8910, Log Rank; Two-sided significance level = 0.05; Hazard Ratio (HR) = 1.03, 95% CI 2-sided [0.64 to 1.68] — Reference level = Chemoradiation

3. Secondary Outcome: Percentage of Participants With Local-regional Progression
Description: Local-regional progression (LRP) is defined as progression within the planned treatment volume (PTV) or outside the PTV but within the same lobe(s) of the lung as the primary tumor or in regional lymph nodes. Progression is defined as change in a known lesion(s) meeting one of the following criteria: [1] ≥ 20% increase in the sum of the longest diameter of target lesions such that the absolute increase must be > 5 mm. [2] Appearance of ≥1 new lesions. LRP time is defined as time from randomization to the date of first LRP, death without LRP (competing risk), or last known follow-up (censored). LRP rates are estimated using the cumulative incidence method. The protocol specifies that the distributions of failure times be compared between the arms, which is reported in the statistical analysis results. One-year rates are provided. Analysis occurred after 102 LRP events were reported.
Time Frame: From randomization to last follow-up. Maximum follow-up at time of analysis was 47.2 months.
Population: Eligible participants
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Chemoradiation | Metformin + Chemoradiation
Number analyzed (Participants) | 81 | 86
percentage of participants | 17.2 [9.7 to 26.6] | 20.5 [12.4 to 30.2]
Statistical Analysis 1: Comparison: Chemoradiation vs Metformin + Chemoradiation; Test type: Superiority; p = 0.4075, Log Rank; Two-side significance level = 0.05; Hazard Ratio (HR) = 1.29, 95% CI 2-sided [0.71 to 2.34] — Reference level = Chemoradiation

4. Secondary Outcome: Percentage of Participants With Distant Metastases
Description: Distant metastasis (DM) is defined as the appearance of ≥ 1 new lesions at any site (including pleural or pericardial effusion) outside of the following: the planned treatment volume, the same lobe(s) of the lung as the primary tumor, or regional lymph nodes. Time to DM is defined as time from randomization to the date of first DM, death without DM (competing risk), or last known follow-up (censored). DM rates are estimated using the cumulative incidence method. The protocol specifies that the distributions of failure times be compared between the arms, which is reported in the statistical analysis results. One-year rates are provided. Analysis occurred after 102 progression-free survival events were reported.
Time Frame: From randomization to last follow-up. Maximum follow-up at time of analysis was 47.2 months.
Population: Eligible participants
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Chemoradiation | Metformin + Chemoradiation
Number analyzed (Participants) | 81 | 86
percentage of participants | 17.2 [9.7 to 26.6] | 20.5 [12.4 to 30.2]
Statistical Analysis 1: Comparison: Chemoradiation vs Metformin + Chemoradiation; Test type: Superiority; p = 0.4075, Log Rank; Two-sided significance level = 0.05; Hazard Ratio (HR) = 1.29, 95% CI 2-sided [0.71 to 2.34] — Reference level = Chemoradiation

5. Secondary Outcome: Percentage of Participants With Treatment-related Grade 3 or Higher Adverse Events
Description: Adverse events (AE) were graded using the Common Terminology Criteria for Adverse Events (CTCAE) v4.0. Grade refers to the severity of the AE. The CTCAE v4.0 assigns Grades 1 through 5 with unique clinical descriptions of severity for each AE based on this general guideline: Grade 1 Mild, Grade 2 Moderate, Grade 3 Severe, Grade 4 Life-threatening or disabling, Grade 5 Death related to adverse event. "Treatment-related" is defined definitely, probably, or possibly related to treatment.
Time Frame: From start of treatment to last follow-up. Maximum follow-up at time of analysis was 47.2 months.
Population: Eligible participants who started protocol treatment
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Chemoradiation | Metformin + Chemoradiation
Number analyzed (Participants) | 76 | 82
percentage of participants | 67.1 [55.4 to 77.5] | 63.4 [52.1 to 73.8]
Statistical Analysis 1: Comparison: Chemoradiation vs Metformin + Chemoradiation; Test type: Superiority; p = 0.6266, Chi-squared; Two-sided significance level = 0.05; Odds Ratio (OR) = 0.92, 95% CI 2-sided [0.47 to 1.80] — Reference level = Chemoradiation

ADVERSE EVENTS:
Time Frame: Adverse events were to be reported weekly during dose escalation on metformin arm, end of chemoradiation, end of post-radiation chemotherapy/metformin, 4-6 weeks follow-up, every 3 months for 2 years follow-up, every 6 months through 5 years follow-up, yearly until study termination completion.
Arm/Group | Chemoradiation | Metformin + Chemoradiation
All-Cause Mortality (participants affected / at risk) | 31/76 | 34/82
Serious Adverse Events (participants affected / at risk) | 31/76 | 27/82
Other Adverse Events (participants affected / at risk) | 75/76 | 79/82
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Chemoradiation (N=76) | Metformin + Chemoradiation (N=82)
Anemia (Blood and lymphatic system disorders) | 3 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 4 | 0
Atrial fibrillation (Cardiac disorders) | 2 | 1
Atrial flutter (Cardiac disorders) | 0 | 1
Cardiac disorders - Other (Cardiac disorders) | 1 | 0
Heart failure (Cardiac disorders) | 1 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 1
Diarrhea (Gastrointestinal disorders) | 1 | 0
Dysphagia (Gastrointestinal disorders) | 2 | 0
Esophageal pain (Gastrointestinal disorders) | 1 | 1
Esophagitis (Gastrointestinal disorders) | 4 | 5
Mucositis oral (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0
Death NOS (General disorders) | 2 | 0
Fatigue (General disorders) | 1 | 2
Fever (General disorders) | 0 | 1
Infusion related reaction (General disorders) | 2 | 1
Malaise (General disorders) | 0 | 1
Endocarditis infective (Infections and infestations) | 1 | 0
Esophageal infection (Infections and infestations) | 1 | 0
Infections and infestations - Other (Infections and infestations) | 0 | 2
Lung infection (Infections and infestations) | 5 | 6
Pleural infection (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 1 | 2
Urinary tract infection (Infections and infestations) | 1 | 0
Dermatitis radiation (Injury, poisoning and procedural complications) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1
Spinal fracture (Injury, poisoning and procedural complications) | 0 | 1
Investigations - Other (Investigations) | 1 | 0
Lymphocyte count decreased (Investigations) | 3 | 1
Neutrophil count decreased (Investigations) | 5 | 3
Platelet count decreased (Investigations) | 4 | 1
Weight loss (Investigations) | 0 | 1
White blood cell decreased (Investigations) | 4 | 2
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Hypercalcemia (Metabolism and nutrition disorders) | 0 | 1
Hypokalemia (Metabolism and nutrition disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 2
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 | 2
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Intracranial hemorrhage (Nervous system disorders) | 1 | 0
Peripheral motor neuropathy (Nervous system disorders) | 1 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 1 | 0
Presyncope (Nervous system disorders) | 1 | 0
Reversible posterior leukoencephalopathy syndrome (Nervous system disorders) | 0 | 1
Seizure (Nervous system disorders) | 1 | 0
Stroke (Nervous system disorders) | 1 | 1
Syncope (Nervous system disorders) | 0 | 2
Tremor (Nervous system disorders) | 0 | 1
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 5 | 5
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 3 | 2
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Respiratory, thoracic and mediastinal disorders - Other (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Thromboembolic event (Vascular disorders) | 1 | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Chemoradiation (N=76) | Metformin + Chemoradiation (N=82)
Anemia (Blood and lymphatic system disorders) | 50 | 46
Atrial fibrillation (Cardiac disorders) | 2 | 5
Sinus tachycardia (Cardiac disorders) | 3 | 7
Hearing impaired (Ear and labyrinth disorders) | 5 | 1
Blurred vision (Eye disorders) | 4 | 4
Abdominal pain (Gastrointestinal disorders) | 6 | 4
Constipation (Gastrointestinal disorders) | 35 | 29
Diarrhea (Gastrointestinal disorders) | 25 | 46
Dry mouth (Gastrointestinal disorders) | 6 | 7
Dyspepsia (Gastrointestinal disorders) | 11 | 15
Dysphagia (Gastrointestinal disorders) | 31 | 29
Esophageal pain (Gastrointestinal disorders) | 5 | 9
Esophagitis (Gastrointestinal disorders) | 29 | 37
Flatulence (Gastrointestinal disorders) | 2 | 5
Gastroesophageal reflux disease (Gastrointestinal disorders) | 4 | 10
Gastrointestinal disorders - Other (Gastrointestinal disorders) | 2 | 5
Mucositis oral (Gastrointestinal disorders) | 9 | 4
Nausea (Gastrointestinal disorders) | 43 | 48
Vomiting (Gastrointestinal disorders) | 18 | 34
Chills (General disorders) | 4 | 8
Edema limbs (General disorders) | 9 | 9
Fatigue (General disorders) | 61 | 66
Fever (General disorders) | 11 | 13
Infusion related reaction (General disorders) | 4 | 6
Localized edema (General disorders) | 4 | 2
Non-cardiac chest pain (General disorders) | 13 | 15
Pain (General disorders) | 21 | 21
Bronchial infection (Infections and infestations) | 5 | 2
Infections and infestations - Other (Infections and infestations) | 7 | 3
Lung infection (Infections and infestations) | 4 | 7
Skin infection (Infections and infestations) | 4 | 1
Upper respiratory infection (Infections and infestations) | 8 | 7
Urinary tract infection (Infections and infestations) | 5 | 4
Dermatitis radiation (Injury, poisoning and procedural complications) | 15 | 19
Fall (Injury, poisoning and procedural complications) | 4 | 7
Alanine aminotransferase increased (Investigations) | 10 | 7
Alkaline phosphatase increased (Investigations) | 13 | 9
Aspartate aminotransferase increased (Investigations) | 10 | 4
Blood bilirubin increased (Investigations) | 4 | 3
Creatinine increased (Investigations) | 9 | 7
Lymphocyte count decreased (Investigations) | 35 | 32
Neutrophil count decreased (Investigations) | 21 | 31
Platelet count decreased (Investigations) | 36 | 37
Weight gain (Investigations) | 4 | 3
Weight loss (Investigations) | 19 | 30
White blood cell decreased (Investigations) | 40 | 39
Anorexia (Metabolism and nutrition disorders) | 19 | 33
Dehydration (Metabolism and nutrition disorders) | 15 | 18
Hyperglycemia (Metabolism and nutrition disorders) | 14 | 23
Hypernatremia (Metabolism and nutrition disorders) | 5 | 2
Hypoalbuminemia (Metabolism and nutrition disorders) | 25 | 21
Hypocalcemia (Metabolism and nutrition disorders) | 10 | 10
Hypokalemia (Metabolism and nutrition disorders) | 14 | 16
Hypomagnesemia (Metabolism and nutrition disorders) | 9 | 16
Hyponatremia (Metabolism and nutrition disorders) | 15 | 24
Arthralgia (Musculoskeletal and connective tissue disorders) | 13 | 7
Back pain (Musculoskeletal and connective tissue disorders) | 13 | 12
Bone pain (Musculoskeletal and connective tissue disorders) | 4 | 4
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 17 | 19
Musculoskeletal and connective tissue disorder - Other (Musculoskeletal and connective tissue disorders) | 4 | 4
Myalgia (Musculoskeletal and connective tissue disorders) | 14 | 16
Pain in extremity (Musculoskeletal and connective tissue disorders) | 7 | 10
Dizziness (Nervous system disorders) | 16 | 19
Dysgeusia (Nervous system disorders) | 14 | 16
Headache (Nervous system disorders) | 8 | 23
Paresthesia (Nervous system disorders) | 8 | 6
Peripheral motor neuropathy (Nervous system disorders) | 4 | 2
Peripheral sensory neuropathy (Nervous system disorders) | 31 | 35
Anxiety (Psychiatric disorders) | 12 | 9
Confusion (Psychiatric disorders) | 5 | 6
Depression (Psychiatric disorders) | 8 | 4
Insomnia (Psychiatric disorders) | 13 | 13
Cough (Respiratory, thoracic and mediastinal disorders) | 45 | 40
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 42 | 42
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 5 | 7
Hiccups (Respiratory, thoracic and mediastinal disorders) | 2 | 6
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 4 | 10
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 9 | 5
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 8 | 6
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 16 | 14
Productive cough (Respiratory, thoracic and mediastinal disorders) | 11 | 11
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 5 | 4
Respiratory, thoracic and mediastinal disorders - Other (Respiratory, thoracic and mediastinal disorders) | 9 | 7
Sore throat (Respiratory, thoracic and mediastinal disorders) | 12 | 9
Wheezing (Respiratory, thoracic and mediastinal disorders) | 9 | 6
Alopecia (Skin and subcutaneous tissue disorders) | 28 | 28
Dry skin (Skin and subcutaneous tissue disorders) | 5 | 6
Pruritus (Skin and subcutaneous tissue disorders) | 4 | 6
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 10 | 5
Skin and subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 4 | 8
Hot flashes (Vascular disorders) | 6 | 4
Hypertension (Vascular disorders) | 9 | 14
Hypotension (Vascular disorders) | 11 | 11
Thromboembolic event (Vascular disorders) | 3 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI's are required to abide by the sponsor's publication guidelines which require review by coauthors and subsequent review and approval by the sponsor.

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-11-01): https://cdn.clinicaltrials.gov/large-docs/47/NCT02186847/Prot_SAP_001.pdf
  • Informed Consent Form (2018-11-01): https://cdn.clinicaltrials.gov/large-docs/47/NCT02186847/ICF_000.pdf